CLINICAL TRIAL: NCT02192073
Title: Prospective Analysis of Arthroscopic Suprapectoral and Open Subpectoral Biceps Tenodesis: 1 Year Follow-Up
Brief Title: Analysis of Suprapectoral and Subpectoral Biceps Tenodesis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Carla Edwards, Clinical Research Manger, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13081402
Record Dates: First submitted 2014-05-21; First posted 2014-07-16 (Estimated); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Biceps Tendonitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Suprapectoral Biceps Tenodesis (Active Comparator): Suprapectoral Biceps Tenodesis involves detaching the long head of biceps from it's origin and reattaching it to humerus in the superior border of the pectoralis major insertion
  Interventions: Procedure: Suprapectoral Biceps tenodesis
- Subpectoral Biceps Tenodesis (Active Comparator): Subpectoral Biceps Tenodesis involves detaching the long head of biceps from it's origin and reattaching it to humerus in the inferior border of the pectoralis major insertion
  Interventions: Procedure: Subpectoral biceps tenodesis

INTERVENTIONS:
Procedure: Suprapectoral Biceps tenodesis
  Arms: Suprapectoral Biceps Tenodesis
Procedure: Subpectoral biceps tenodesis
  Arms: Subpectoral Biceps Tenodesis

SUMMARY:
Biceps pathology typically includes pain in the anterior shoulder that is reproduced with provocative maneuvers. However, optimal treatment of patient with this diagnosis is not clear and can include tenotomy (cutting the biceps) or various forms of tenodesis (cutting then reattaching). As tenotomy can lead to cosmetic deformity and anterior humeral discomfort from spasms, many surgeons perform tenodesis. There are various techniques for tenodesis. This study will compare 2 methods: suprapectoral (doing the surgery using an incision higher in the shoulder) versus subpectoral fixation (surgery which involves making an incision lower in the shoulder).

Purpose of the study is to prospectively determine whether arthroscopic suprapectoral or open subpectoral biceps tenodesis results in better function.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo biceps tenodesis
* Pain at intertubercular groove
* Anterior Humeral pain
* Patient agrees to follow up and consent

Exclusion Criteria:

* Biceps Tenotomy
* Revision biceps procedure
* Prior SLAP or labral repair
* Concomitant subscapularis repair
* More than 1 rotator cuff repair at time of surgery
* Concomitant arthroplasty
* Prior infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2018-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
American Shoulder and Elbow Surgeons (ASES) Shoulder Score | 1 year
  Validated outcome score assessing pain and function of shoulder

SECONDARY OUTCOMES:
Constant Score | 1 year
  Validated score to assess shoulder pain and function

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil N Verma, MD, Principal Investigator — Rush Univeristy Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Forsythe B, Berlinberg EJ, Diaz CC, Korrapati A, Agarwalla A, Patel HH, Cole BJ, Cvetanovich GL, Yanke AB, Romeo AA, Verma NN. No Difference in Clinical Outcomes for Arthroscopic Suprapectoral Versus Open Subpectoral Biceps Tenodesis at Midterm Follow-up: A Randomized Prospective Analysis. Am J Sports Med. 2022 May;50(6):1486-1494. doi: 10.1177/03635465221084731. PMID 35507468